CLINICAL TRIAL: NCT00950144
Title: Illness Perception, Pain and Symptom Distress in Gastrointestinal Cancers
Brief Title: Studying Pain and Symptom Distress in Patients With Advanced Colon Cancer, Rectal Cancer, Pancreatic Cancer, or Liver Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Virginia Sun, City of Hope Comprehensive Cancer Center
Other Study IDs: 08131; P30CA033572 (NIH); CHNMC-08131; CDR0000632905 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer; Depression; Fatigue; Liver Cancer; Pain; Pancreatic Cancer
Keywords: pain; depression; fatigue; stage III colon cancer; stage IV colon cancer; recurrent colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Colorectal Neoplasms; Depression; Fatigue; Liver Neoplasms; Pain; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying a patient's understanding of his or her illness, pain, symptoms, and quality-of-life may help the study of advanced cancer and may help patients live more comfortably.

PURPOSE: This clinical trial is studying pain and symptom distress in patients with advanced colon cancer, rectal cancer, pancreatic cancer, or liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe illness perception as indicated in the five domains of the Common Sense Model (i.e., identity, cause, time line, consequences, controllability) and their relationship to symptom distress in patients with colon, rectal, pancreatic, or liver (i.e., hepatocellular carcinoma) cancer.
* To describe pain and other symptoms and their relationship to overall symptom distress in these patients.
* To describe overall quality of life (QOL) and its specific summary scales in these patients.
* To explore the relationship among characteristics (i.e., sociodemographic, disease, health status) associated with illness perceptions, overall symptom distress, and QOL in these patients.

OUTLINE: Patients undergo an empirical examination of illness perceptions as predictors of disease, specifically from the five domains in the Common Sense Model. Patients undergo an assessment of the relationship between influencing characteristics (i.e., sociodemographic), symptoms, and behavioral factors (i.e., illness perceptions, overall symptom distress, and quality of life). Patients complete questionnaires to evaluate demographics by the Sociodemographic, Disease, and Health Status Tool; illness perception by the Illness Perception Questionnaire-Revised (IPQ-R); symptoms and symptom distress by the Memorial Symptom Assessment Scale (MSAS) and Brief Pain Inventory; and quality of life by the SF-12. Patients also undergo a medical chart review and self-report on sociodemographic characteristics.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colon, rectal, pancreatic, or liver (i.e., hepatocellular carcinoma) cancer

  * Stage III or IV colon, rectal, or pancreatic cancer
  * Child-Pugh class B or C hepatocellular carcinoma

PATIENT CHARACTERISTICS:

* Able to read English
* Able to provide written informed consent and complete questionnaire packet

PRIOR CONCURRENT THERAPY:

* Any treatment modality (e.g., chemotherapy, radiotherapy, surgery) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at the City of Hope Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Illness perception as indicated in the five domains of the Common Sense Model (i.e., identity, cause, time line, consequences, controllability) and their relationship to symptom distress | At study entry
Pain and other symptoms, and their relationship to overall symptom distress | At study entry
Overall quality of life (QOL) and its specific summary scales | At study entry
Relationship among characteristics (i.e., sociodemographic, disease, health status) associated with illness perceptions, overall symptom distress, and QOL) | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, RN, MSN, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States